CLINICAL TRIAL: NCT04244721
Title: Effectiveness of PACT Intervention, Delivered by Parents, Guided by Videoconference, on the Autism of Their Children With ASD
Brief Title: Effectiveness of a Parent-mediated Intervention With PACT on Children With ASD
Acronym: IFPAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-A02516-49
Record Dates: First submitted 2020-01-21; First posted 2020-01-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder
Keywords: interventions Early Start Denver Model (ESDM); Preschool Autism Communication Therapy (PACT)
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: To make the comparison between the two groups on autism symptoms outcome measured with ADOS-2, with a power of 80% and an improvement of 0.6 points, we need 198 children (99 per group). After taking into account of a 20% consensual withdrawals and poor compliance with PACT, 238 children (119 per group) will be required. Each center will therefore have to include 50 children during the inclusion period.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a group of children receiving the usual therapy (TAU) (Sham Comparator): Children will receive therapies available in the community as speech language therapist or occupational therapist.
  Interventions: Other: Treatment As Usual (TAU)
- a group of children receiving TAU plus the PACT intervention. (Experimental): Professionals guide parents in the PACT therapy by videoconference. Sessions between parent and professionals are every 15 days for 6 months. Each session lasts one hour. At the end of the 12 sessions, additional booster sessions (one session per month over 6 months) will allow parents to maintain their skills. Parents will use therapy with their children in daily home practice. The aims of PACT therapy is to improve synchrony in the communication between the child and the parents. Improvement of the synchrony will mediate the decrease of autism symptoms of the child.
  Interventions: Other: Preschool Autism Communication Therapy (PACT)

INTERVENTIONS:
Other: Preschool Autism Communication Therapy (PACT) — Professionals guide parents in the PACT therapy by videoconference. Sessions between parent and professionals are every 15 days for 6 months. Each session lasts one hour. At the end of the 12 sessions, additional booster sessions (one session per month over 6 months) will allow parents to maintain their skills. Parents will use therapy with their children in daily home practice. The aims of PACT therapy is to improve synchrony in the communication between the child and the parents. Improvement of the synchrony will mediate the decrease of autism symptoms of the child.
  Arms: a group of children receiving TAU plus the PACT intervention.
Other: Treatment As Usual (TAU) — Children will receive therapies available in the community as speech language therapist or occupational therapist.
  Arms: a group of children receiving the usual therapy (TAU)

SUMMARY:
Autism Spectrum Disorder (ASD) is a neuro-developmental disorders. There are different types of interventions. Among these interventions Early Start Denver Model (ESDM) and Preschool Autism Communication Therapy (PACT) have proved efficacy at short and long term. PACT is the therapy with the highest evidences when Parents delivered the intervention themselves.

DETAILED DESCRIPTION:
In PACT, parents are guided, generally in face to face, by a professional to improve the synchrony and communication with their children with ASD. Then, it is recommended to the parents to practice the therapy daily at home. In France, this type of early intervention is poorly developed and is only accessible in specialized centers located in large urban centers. Guiding parents by videoconferencing could make this intervention accessible to families in undeserved areas. The objective of this study is to evaluate the effectiveness of a PACT intervention delivered by parents and guided by videoconferencing, on the autism in their children with ASD, aged 18 to 36 months at the inclusion.

This is a mixed (quantitative and qualitative), multicenter, controlled, randomized, open-label study, comparing a group of children receiving usual care and one of whose parents is trained and accompanied by videoconferencing to developmental techniques as described in the PACT, to a group of children benefiting only from the usual care provided by the community. The primary endpoint was the severity of autism measured with the ADOS-2 (2012 Autism Diagnostic Observation Schedule) severity score (CSS) at 12 months. A total of 212 children will be included in the study (106 / group).

ELIGIBILITY:
Inclusion Criteria:

Child with autism Spectrum disorder

* Symptoms in autism with a severity superior to 4 as measure by ADOS-2
* Positive ADI (Autism Diagnostic Interview)
* Diagnostic done by a multidisciplinary team
* Nonverbal IQ above 12 months Having health assurance

Exclusion Criteria:

For the child

* Child with a twin brother or sister with ASD or having a brother or sister already included in this study
* Epilepsy requiring medication
* Severe hearing or visual impairment
* Identification of a genetic anomaly causes participation in the intervention or validity of the data (determined by the principal investigator on a case-by-case basis)

For the parents

* Severe hearing or visual impairment
* Severe psychiatric disorder
* Unstable somatic disorders preventing intervention
* Lack of Internet access
* Parent not available for regular follow-up
* Opposition of one parent to the child's participation in a study
* Already receiving PACT therapy or any other intensive intervention (e.g. Denver)

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 212 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Autism severity | 12 months
  Change between baseline and 12 months in the overall raw score at ADOS-2 (Autism Diagnostic Observation Schedule version 2), Module 1

SECONDARY OUTCOMES:
Social Interactions of the child | 6 and 12 months
  Social Interactions measured with the total score of the BOSCC (Brief Observation of Social Communication Change).
  The test contains 9 items that are meant to capture the quality of a child's social interaction, for which the total scores ranges from 0 to 45, and 3 items describing restricted a repetitive behavior, which is also part of the ASD symptomatology, the total score of which ranges from 0 to 15. Three additional items are coded to add information on symptoms that might be present although they are not specifically part of the ASD syndrome, and refer to activity level, disruptive behavior, and anxious behaviors. The BOSCC total score consists in the sum of the total score obtained in the first twelve items (ASD specific symptoms), and ranges from 0 to 60, with the three extra items added separately to integrate information. In the total and subscale scores, higher scores correspond to more severe symptoms.
Parent-child synchrony and initiative in communication | 6 and 12 months
  Parent-child synchrony and initiative in communication measure with DCMA (Dyadic Communication Measure for autism)
Number of words produced by the child | 12 months
  Number of words produced by the child measured with global score of the french scale " Développement du Langage de Production en Français " (DLPF)
Number of words produced by the child | 12 months
  Number of words produced by the child measured with global score of the Mullen Scale of early learning (MSEL)
Adaptative behavior | 12 months
  Adaptative behavior measured with VABS (Vineland Adaptative Behaviour Scales 2).
  The Vineland Adaptive Behavior Scales (VABS; Sparrow et al., 1984) comprises four domains, that is, communication, daily living skills, socialization and motor skills, for assessing adaptive functioning in children aged 3 to 12 years old. The raw score in each domain and total raw score are converted to an age-equivalent score. The domain scores are also expressed as standard scores with a mean of 100 and standard deviation of 15. The range for each subscale is from 20 to 140. The subscales are summed to compute a total score, ranging from 80 to 560. The higher the scores are, the better adaptive functioning the children achieve.
Autism Family Experience | 12 months
  Measured with the questionnaire Autism Family Experience. The Autism Family Experience Questionnaire (AFEQ) is a parent/Caregiver form used to measure impact of autism interventions on family experience and quality of life. The AFEQ included both positively and negatively worded statements and is scored on an order scale: 1 = always to 5 = never, with an option for "Not Applicable". 4 domains are evaluated : experience of being a parent, family life, child development understanding and social relationships, child symptoms.A higher score means a worse outcome.
Characteristics of the parents | 12 months
  Measured with General Health Questionnaire (GHQ-28). The GHQ-28 is a 28-item self-report used to psychological stress. The GHQ focuses on two main classes of phenomena: 1) inability to carry out one's normal healthy functions; and 2) emergence of new phenomena that are distressing.
  It consists of 28 items, divided into 4 sub-scales. It contains 4 sub-scales: A (somatic symptoms), B (anxiety/insomnia), C (social dysfunction), and D (severe depression). There are 4 possible answers to each question. The Likert scoring system assigns a value from 0 to 3 to each of the 4 possible answers. A higher score means a worse outcome.
Characteristics of the parents | 12 months
  Measured with ISP (Indice of Parental Stress). A self-report inventory designed to measure the overall level of parenting stress an individual is experiencing and it examine stressors associated specifically with the parental role and do not include stresses associated with other life roles and events. The PSI-SR has strong psychometric properties and has been used in a number of studies of autism and parent training. It contains 36 items, each rated on a five-point Likert scale (1-5), with higher scores indicative of more parenting stress and includes Parental Distress (PD), Parent-Child Dysfunctional Interaction (P-CDI) and Difficult Child (DC) sub-scales.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jurek L, Occelli P, Denis A, Amestoy A, Maffre T, Dauchez T, Oreve MJ, Baghdadli A, Schroder C, Jay A, Zelmar A, Revah-Levy A, Gallifet N, Aldred C, Garg S, Green J, Touzet S, Geoffray MM; IFPAD study group. Efficacy of parent-mediated communication-focused treatment in toddlers with autism (PACT) delivered via videoconferencing: a randomised controlled trial study protocol. BMJ Open. 2021 Apr 7;11(4):e044669. doi: 10.1136/bmjopen-2020-044669. PMID 33827837